CLINICAL TRIAL: NCT03681054
Title: Effects of Guided Dietary Patterns on Metabolic Outcomes in Overweight Pregnant Women With Gestational Diabetes and on Offspring Body Composition
Brief Title: Dietary Management of Gestational Diabetes
Acronym: eMOM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); Aalto University (Other); Finnish Institute for Health and Welfare (Other Government); City of Helsinki (Other); UKK Institute (Other)
Responsible Party: Principal Investigator, Saila Koivusalo, Principal Investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUS/1792/2016_2
Record Dates: First submitted 2018-09-20; First posted 2018-09-21 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Diabetes, Gestational; Dietary Modification; Glucose Intolerance During Pregnancy; Body Composition; Birth Weight
Keywords: Nutrition; Dietary Counseling; Diet; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Birth Weight | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbohydrate restricted diet (Experimental): Dietary intervention: moderately carbohydrate restricted diet. Parallel phase starts after study period I and the diet is followed until labor.
  Interventions: Other: Carbohydrate restricted diet
- Plant-protein based diet (Experimental): Dietary intervention: plant-protein based diet, en emphasis on healthy Nordic foods. Parallel phase starts after study period I and the diet is followed until labor.
  Interventions: Other: Plant-protein based diet

INTERVENTIONS:
Other: Carbohydrate restricted diet — The intervention is implemented by individual face-to-face counseling and mobile-phone counseling by a nutritionist, as well as food bags and recipes suitable for the diet. Targets: fruits and vegetables 500 g/d, fish 2 times/wk, low-fat instead of high-fat meat, red meat ≤ 3 times/wk, low-fat instead of high-fat dairy, high-fibre instead of low-fibre grains, vegetable oils (excluding palm oil and coconut oil) and soft margarine instead of animal fats, moderate reduction of carbohydrates (targets for macronutrients: carbohydrates 40 E%; fat 40 E%; protein 20 E%; dietary fiber 32g, energy intake approximately 2000 kcal/d; protein intake 20 E%; sucrose: <10 E%; fatty acids: saturated fatty acids < 10 E%, polyunsaturated fatty acids 5-10 E% and the rest of fat as monounsaturated fatty acids)
  Arms: Carbohydrate restricted diet
Other: Plant-protein based diet — The intervention is implemented by individual face-to-face counseling and mobile-phone counseling by a nutritionist, as well as food bags and recipes suitable for the diet. Targets: fruits and vegetables 1 kg/d; fish 3/wk; high-fibre grains, mainly rye, oat and barley; plant protein instead of meat protein; low-fat fermented dairy instead of other dairy; rapeseed oil and rapeseed-based margarine instead of other fats; no carbohydrate restriction (targets for macronutrients: carbohydrates 50 E%; fat 30 E%; protein 20 E%; dietary fiber 36g, energy intake approximately 2000 kcal/d; protein intake 20 E%; sucrose: <10 E%; fatty acids: saturated fatty acids < 10 E%, polyunsaturated fatty acids 5-10 E% and the rest of fat as monounsaturated fatty acids)
  Arms: Plant-protein based diet

SUMMARY:
eMOM is a randomized, controlled trial to compare the effects of two different dietary interventions during pregnancy. The comparison is based on tissue glucose content (using continuous glucose monitoring system) in pregnant women and on neonate body composition. The recruited women (n=60) have been diagnosed with gestational diabetes mellitus, and are of Caucasian origin. Of the study diets, one is moderately carbohydrate restricted and the other one is high on plant-based protein with an emphasis on healthy Nordic foods. The study has two two-week study periods that are carried out on approximately gestational weeks 24-28 (period I) and 34-36 (period II). Continuous glucose monitoring and other measurements (accelerometer, 3-day food record, gut microbiota, serum lipids, metabolomics, epigenetics etc.) are done during these study periods. At the beginning of the study, before study period I, the participants are randomized to either one of the intervention diets. The first study period consists of a crossover phase in which the participants receive three days' worth of food according to one of the intervention diets (according to the randomization) after which there is a three-day wash-out period. After the wash-out period, the participants receive three days' worth of food according to the other diet. After the first study period, a nutritionist advises the lastly followed intervention diet to the participant and the diet is followed until delivery. To ensure the diet is followed, the participants gets at least three personal face-to-face counseling sessions, phone calls, mobile reminders, recipes and food items. After delivery, the infant's body composition, epigenetic markers of cord blood and placenta, gut microbiome and urine metabolomics are measured.

ELIGIBILITY:
Inclusion Criteria:

- Gestational diabetes at enrollment

Exclusion Criteria:

* Gestational weeks exceed 28+6
* Multiple pregnancy
* Food allergies or restrictions (other than lactose intolerance)
* Mother's or father's ethnic background other than Caucasian
* Type 1 or type 2 diabetes
* Medication which affects glucose metabolism
* Cholesterol medication
* Drug or alcohol abuse
* Psychiatric illness which affects participation in the study
* Factors hampering communication (e.g. lack of Finnish skills)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Mother: The percentage of time spent within the gestational diabetes glucose target range (<7,8 mmol/l) in cross-over phase | Study period I: during a 3 day intervention-diet period within gestational weeks 24-28
  Measured with FreeStyle®Libre, Continuous Glucose Monitoring system
Mother: The percentage of time spent within the gestational diabetes glucose target range (<7,8 mmol/l) | Study period II: during a 14 day period within gestational weeks 34-36
  Measured with FreeStyle®Libre, Continuous Glucose Monitoring system
Child: Neonatal body fat% | one measure within 0-2 days after birth of the child
  Neonatal body fat%; Measured with PEA POD Cosmed® Infant Body Composition Assessment system

SECONDARY OUTCOMES:
Mother: Glycaemic variability in crossover phase | Study period I: during a 3 day intervention-diet period within gestational weeks 24-28
  Measured with FreeStyle®Libre, Continuous Glucose Monitoring system
Mother: Glycaemic variability | Study period II: during a 14 day period within gestational weeks 34-36
  Measured with FreeStyle®Libre, Continuous Glucose Monitoring system
Percentage of participants on GDM medication | Up to 42 gestational weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seppo Heinonen, prof, Study Director — Head of department of obs and gyn/Helsinki University Hospital
Locations (1):
- Helsinki university central hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Markussen LT, Kivela J, Lindstrom J, Ollikainen M, Kyto M, Heinonen S, Koivusalo S, Meinila J. Glycemic control in women with GDM: insights from a randomized controlled pilot trial on plant-based Nordic healthy diet versus moderately carbohydrate restricted diet. BMC Nutr. 2025 Jan 16;11(1):12. doi: 10.1186/s40795-024-00988-x. PMID 39815337
- [Derived] Markussen LT, Kivela J, Lindstrom J, Ashrafi RA, Heinonen S, Koivusalo S, Meinila J. Short-term effect of plant-based Nordic diet versus carbohydrate-restricted diet on glucose levels in gestational diabetes - the eMOM pilot study. BMC Nutr. 2023 Jul 14;9(1):87. doi: 10.1186/s40795-023-00744-7. PMID 37452403